CLINICAL TRIAL: NCT03339479
Title: Dielectric Property Test Compared With Frozen Pathological Section in the Rapid Diagnosis of Lung Nodules/Mass: a Diagnostic Clinical Trial
Brief Title: Dielectric Property Test Compared With Frozen Pathological Section in the Rapid Diagnosis of Lung Nodules/Mass
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NFEC-2017-070
Record Dates: First submitted 2017-08-21; First posted 2017-11-13 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-05

CONDITIONS: Lung Nodules; Lung Mass
Keywords: dielectric property; lung nodules; differential diagnosis; frozen pathological examination

STUDY DESIGN:
Intervention Model Description: self-control method
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- dielectric property test (Experimental): The patient with lung nodules/mass is firstly arranged to be tested for dielectric property after the nodules/mass resection and cutting open.
  Interventions: Diagnostic Test: dielectric property test
- frozen pathological examination (Placebo Comparator): The resected lung nodules/mass will be sent for frozen pathological examination after dielectric property test.
  Interventions: Diagnostic Test: frozen pathological examination
- final pathological examination (Other): The resected lung nodules/mass will undergo the final pathological examination for final diagnosis after dielectric property test and frozen pathological examination.
  Interventions: Diagnostic Test: final pathological examination

INTERVENTIONS:
Diagnostic Test: dielectric property test — Test the dielectric property of resected lung nodules/mass through a touching probe after the lung tissue with nodules/mass has been resected and cut open, which usually takes only 1-5 minutes.
  Arms: dielectric property test
Diagnostic Test: frozen pathological examination — And after the dielectric property test, the lung tissue will be sent for frozen pathological examination.
  Arms: frozen pathological examination
Diagnostic Test: final pathological examination — All of the lung nodules/mass will be diagnosed by final pathological examination and recognized as the final diagnosis after surgery.
  Arms: final pathological examination

SUMMARY:
Patients with lung nodules/mass found by CT (computed tomography) or PET (positron emission tomography) who agree to receive lung resection are arranged to test the dielectric property before receiving the frozen pathological examination. And the final pathological results are recognized as the standard diagnosis. Then the sensitivity and specificity of the dielectric property test will be evaluated comparing with the frozen pathological examination.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lung nodules/mass found by CT or PET who agree to receive lung resection;
* Diameter of the lung nodule/mass is longer than 8 millimeters;
* More than 50% of the lung nodule/mass is solid component by image examination;
* Diameter of the solid component is longer than 5 millimeters by intraoperative exploration.

Exclusion Criteria:

* Cutting open the resected nodule/mass will interfered with the pathological examination;
* Diameter of the solid component is shorter than 5 millimeters by intraoperative cutting open;
* Cutting open the lung nodule/mass will cause great damage to the patient, such as inducing allergic shock.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Estimated)
Dates: Start 2017-05-25 (Actual); Primary Completion 2020-05-24 (Estimated); Study Completion 2020-05-24 (Estimated)

PRIMARY OUTCOMES:
sensitivity of dielectric property test in diagnosing lung nodules/masses | 3-5 years
  true positive rate in diagnosing lung nodules/masses
specificity of dielectric property test in diagnosing lung nodules/masses | 3-5 years
  true negative rate in diagnosing lung nodules/masses

CONTACTS AND LOCATIONS:
Overall Officials: Di Lu, MD,PhD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guandong, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
The results of dielectric property test, frozen pathological test and final pathological examination of each individual participant.

REFERENCES:
- [Background] Gabriel C, Gabriel S, Corthout E. The dielectric properties of biological tissues: I. Literature survey. Phys Med Biol. 1996 Nov;41(11):2231-49. doi: 10.1088/0031-9155/41/11/001. PMID 8938024
- [Background] Gabriel S, Lau RW, Gabriel C. The dielectric properties of biological tissues: II. Measurements in the frequency range 10 Hz to 20 GHz. Phys Med Biol. 1996 Nov;41(11):2251-69. doi: 10.1088/0031-9155/41/11/002. PMID 8938025
- [Background] Gabriel S, Lau RW, Gabriel C. The dielectric properties of biological tissues: III. Parametric models for the dielectric spectrum of tissues. Phys Med Biol. 1996 Nov;41(11):2271-93. doi: 10.1088/0031-9155/41/11/003. PMID 8938026
- [Background] Joines WT, Zhang Y, Li C, Jirtle RL. The measured electrical properties of normal and malignant human tissues from 50 to 900 MHz. Med Phys. 1994 Apr;21(4):547-50. doi: 10.1118/1.597312. PMID 8058021
- [Background] Lu Y, Li B, Xu J, Yu J. Dielectric properties of human glioma and surrounding tissue. Int J Hyperthermia. 1992 Nov-Dec;8(6):755-60. doi: 10.3109/02656739209005023. PMID 1479201
- [Background] Surowiec AJ, Stuchly SS, Barr JB, Swarup A. Dielectric properties of breast carcinoma and the surrounding tissues. IEEE Trans Biomed Eng. 1988 Apr;35(4):257-63. doi: 10.1109/10.1374. No abstract available. PMID 2834285
- [Background] Fu F, Xin SX, Chen W. Temperature- and frequency-dependent dielectric properties of biological tissues within the temperature and frequency ranges typically used for magnetic resonance imaging-guided focused ultrasound surgery. Int J Hyperthermia. 2014 Feb;30(1):56-65. doi: 10.3109/02656736.2013.868534. Epub 2014 Jan 13. PMID 24417349